CLINICAL TRIAL: NCT02763449
Title: Appetite and Adiposity Across a Continuum of Activity
Acronym: AAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Robin Shook, Assistant Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AAA-1
Record Dates: First submitted 2016-04-04; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Physical Activity and Sedentary Behavior
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedentary (Experimental): Individuals will reduce their physical activity level for 14-days
  Interventions: Behavioral: Self-monitoing
- Active (Experimental): Individuals will increase their physical activity level for 14-days
  Interventions: Behavioral: Self-monitoing

INTERVENTIONS:
Behavioral: Self-monitoing — Participants will self-monitor their physical activity level via activity monitors

SUMMARY:
The purpose of this study is to understand what happens when someone either becomes more active or more inactive. This study will measure your energy intake, energy expenditure, and body composition under normal conditions, when you become active, and when you become inactive.

ELIGIBILITY:
Inclusion Criteria:

* Men and women

  * Age 25-35 yrs
  * BMI ≥25.0 to <35.0 kg/m2
  * Subjective physical activity (pre run-in): Sedentary for the previous 3 months (< 20min, 3 times/week of structured exercise)
  * Objective physical activity (run-in): daily steps/day >4500 yet <7,000 during 7 day run-in period
  * Weight-stable (± 5%) within the previous 3 months
  * Non-smoking for last year
  * Able to provide own transportation to study visits and intervention
  * Not currently involved in any other research study
  * Willing and able to participate in all aspects of the trial including research testing
  * Willing to give informed consent to participate
  * Able to participate in a moderate physical exercise program

Exclusion Criteria:

* Self-reported significant cardiovascular disease including but not limited to serious arrhythmias, cardiomyopathy, congestive heart failure, myocardial infarction, stroke

  * Other self-reported medical conditions including but not limited to metabolic disorders such as diabetes, chronic or recurrent respiratory conditions, active cancer, musculoskeletal disease interfering with exercise, or any serious medical condition that may affect adherence to the protocol or exercising safely, or be aggravated by exercise
  * Medications known to affect exercise performance or metabolism (e.g. thyroid medication, beta-blockers, or stimulants)
  * Excess caffeine use (> 500mg/day)
  * Restrained eater (>13) on the restraint section of the three-factor eating questionnaire
  * Current or past diagnosis of an eating disorder
  * Any self-reported contraindications to exercise according to the American College of Sports Medicine criteria
  * Pregnant or actively trying to become pregnant
  * Gave birth in the past 12 months or <6 months post-lactation
  * Other medical, psychiatric or behavioral factors that in the judgment of the principal investigator may interfere with study participation or the ability to follow the intervention protocol.
  * Known allergy to the metal nickel
  * Known allergies to pasta or tomato sauce

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Appetite- subjective | 14 days
  Change in appetite will be assessed through subjective ratings of hunger and fullness

SECONDARY OUTCOMES:
Appetite- objective | 14 days
  Change in appetite will be assessed through objective measures of appetite-related hormones

IPD SHARING:
Plan to Share IPD: Undecided